CLINICAL TRIAL: NCT06976398
Title: Investigation of Central Sensitisation in Patients With Chronic Non-spesific Neck Pain
Brief Title: Chronic Neck Pain and Central Sensizitation
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-2281
Record Dates: First submitted 2025-05-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Higher sensitization: It will consist of patients who exceed the cut-off score according to the central sensitization scale score.
- Normal sensitization: It will consist of patients with a central sensitization scale score lower than the cut-off score.

SUMMARY:
Chronic neck pain is one of the musculoskeletal pain problems that can cause chronic disability. It is emphasised that individuals with chronic neck pain have difficulty during different activities in their daily lives, and that this problem is a very common health problem that can lead to disability. In the case of chronic neck pain, changes in the pain threshold cause central sensitisation and individuals become more sensitive to pain stimuli. This situation can affect the processing of proprioceptive information and lead to deterioration in proprioceptive perception. This situation leads to perceptual problems in body and neck awareness. Therefore, examining the relationship between the relevant parameters is important in the rehabilitation process. In this context, the aim of the study is to examine the relationship between body awareness and pain, central sensitisation, disability and proprioception in patients with chronic non-specific neck pain.

DETAILED DESCRIPTION:
Chronic neck pain is a common pain problem related to the musculoskeletal system and can lead to permanent (chronic) disability over time. In approximately 50-85% of individuals with neck pain, complaints do not completely improve despite treatment, causing the pain to become chronic. Individuals with chronic neck pain have difficulty performing various activities in their daily lives, and this negatively affects their quality of life. Proprioceptive feedback in the neck region, that is, sensory information that allows the body to perceive its position in space, is very important for proper control of head and neck movements. However, chronic pain can lead to a condition called central sensitization. In this case, the individual's pain threshold decreases and they become more sensitive to stimuli that would normally not cause pain. This increased sensitivity can make it difficult for the brain to process proprioceptive information correctly, which can lead to impairments in body and neck awareness. Therefore, investigating the relationship between body awareness and pain level, central sensitization, disability status and proprioception in individuals with chronic non-specific neck pain is of great importance in terms of developing an effective rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with chronic non-specific neck pain by a doctor
* Being willing to participate in the study

Exclusion Criteria:

* Having psychological disorders, mental disorders, cancer and severe depression
* Having a history of traumatic injury
* Having a history of primary or metastatic spinal malignancy, spinal fracture
* Having a neurological disease (Hemiplegia, Multiple Sclerosis, Parkinson's, etc.)
* Having been diagnosed with advanced osteoporosis
* Having a history of surgical intervention or acute infection in the cervical region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-specific neck pain will be included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Central sensitization | Baseline
  It will be evaluated with the "Central Sensitization Scale". The scale is scored between 0-100 and 40 points and above is recorded as sensitive.
Pain severity | Baseline
  Pain intensity will be assessed with the Numerical Pain Scale. It is scored between 0-10 and the higher the score, the greater the pain intensity.
Pain threshold | Baseline
  Pain threshold will be assessed with an algometer. An increase in the applied pressure indicates a higher pain threshold.
Neck disability | Baseline
  Neck disability will be evaluated with the index. It varies between 0-50 points and the higher the score, the higher the disability.
Proprioception | Baseline
  Proprioception will be recorded as the degree of deviation with the CROM device. As the degree of deviation increases, proprioception worsens.
Body awareness | Baseline
  Body Awareness Questionnaire (BAF) will be used. It varies between 18-126 points and as the score decreases, awareness decreases.
Neck awareness | Baseline
  It will be assessed with the Fremantle Neck Awareness Questionnaire. It varies between 0-36 and as the score increases, awareness decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Gunes, PhD, Study Director — Karabuk University; Melek Turan, Principal Investigator — Karabuk University; Duygu Çataloluk, Principal Investigator — Karabuk University; Aydın Sinan Apaydın, PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Maas LC, Koke A, Bosscher RJ, Twisk JW, Janssen TW, Peters M. Body Awareness as an Important Target in Multidisciplinary Chronic Pain Treatment: Mediation and Subgroup Analyses. Clin J Pain. 2016 Sep;32(9):763-72. doi: 10.1097/AJP.0000000000000320. PMID 26550959
- [Background] Williams DA. Phenotypic Features of Central Sensitization. J Appl Biobehav Res. 2018 Jun;23(2):e12135. doi: 10.1111/jabr.12135. Epub 2018 Jun 27. PMID 30479469
- [Result] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235